CLINICAL TRIAL: NCT01145092
Title: Effects of Six Months of Moderate Resistance- Versus Endurance-Training on Muscle ATP Synthesis in First-Degree Relatives of Patients With Type 2 Diabetes
Acronym: RECO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landsteiner Institut (Other)
Collaborators: Mein Hanusch-Krankenhaus (Other); Karl-Landsteiner Institute for Endocrinology and Metabolism (Unknown); Medical University of Vienna (Other); Lund University (Other); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Landsteiner Institute, Landsteiner Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P15656
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Type 2 Diabetes Mellitus; Insulin Resistance
Keywords: type 2 diabetes; exercise training; ATP-synthesis; intramyocellular lipids; hepatocellular lipids; first degree relatives of T2DM patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Exercise; Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: exercise training, endurance training — The endurance training group exercised on a cycle ergometer (90% of power output determined at the respiratory compensation point = RCP). The duration of each training unit was increased with time. The resistance group trained on 8 weight machines where the workload gradually increased every 2-3 weeks. At week 13 an additional physical examination, OGTT and spiro-ergometry for adjusting the training were performed.

SUMMARY:
Life style intervention including diet and exercise is the recommended strategy for prevention of type 2 diabetes mellitus (T2DM). First-degree relatives of patients with type 2 diabetes mellitus have an increased risk of insulin resistance and a lifetime risk of developing type 2 diabetes of 40%- 80%. Poor physical fitness is a strong indicator of an increased risk of developing diabetes.

Long-term endurance exercise training has been shown to increase insulin sensitivity in sedentary young and elderly individuals, first degree relatives of patients with Type 2 diabetes, glucose intolerant obese, or Type 2 diabetic humans. In type 2 diabetic patients, non-diabetic individuals with IGT and sedentary adults after exercise training of different intensity, different duration and different frequency an increase of insulin sensitivity was found.

However, despite the vast knowledge concerning beneficial effects physical activity for the prevention of T2DM (and many other chronic metabolic disorders) to date wide ranging strategies have not been realized satisfactory. Regardless of age, ethnicity, sex or health status the lack of time is the primary reason for the failure to exercise on a regular basis (or is stated as primary reason). Therefore the investigators aimed at investigating whether a controlled endurance/resistance training twice a week over 6 month might be beneficial for healthy, non obese, first degree relatives with T2DM. Therefore the investigators measure parameters associated with the prevention of T2DM like insulin sensitivity, flux through fATPase and fCK, intramyocellular and hepatocellular lipids.

ELIGIBILITY:
Inclusion Criteria:

* First degree relatives of type 2 diabetic patients
* Age: 18-50 years
* BMI <30 kg/m2 (due to limited MR diameter)
* Normal routine lab tests (blood cell count, kidney, liver, pancreas, thyroid and neuromuscular function)
* Availability within the local area throughout the study
* Ability to understand and sign the consent forms

Exclusion Criteria:

* Current smoking
* Present drug treatment
* Regular exercise training
* Contraindications for MRS studies: claustrophobia and metalliferous implants
* Pregnancy
* HIV or Hepatitis
* Acute disease 2 weeks previous to the examination
* Heart disease
* Hypertension (RR>140/95)
* Liver disease
* Kidney disease
* Pulmonary disease
* Thyroid disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity
  measured by oral glucose tolerance test

SECONDARY OUTCOMES:
incremental test power, oxygen uptake (VO2 in ml.kg-1.min-1), "aerobic threshold" (RCP= respiratory compensation point)
  This test was performed on an electronically braked cycle ergometer
ATP-Synthesis
  measured with 13C NMR
liver lipid content
  measured with 1H NMR
skeletal muscle lipid content
  measured by 1H NMR

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., Study Director — Institute for Clinical Diabetology, German Diabetes Center (Leibniz Center for Diabetes Research), Department of Metabolic Diseases, Heinrich-Heine University and University Clinics Düsseldorf, Germany
Locations (1):
- Landsteiner Institute, Vienna, Vienna, Austria